CLINICAL TRIAL: NCT05050409
Title: SMART Embedded Intervention for Military Postsurgical Engagement Readiness
Acronym: SEMPER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: The Geneva Foundation (Other)
Responsible Party: Principal Investigator, Eric Garland, Distinguished Professor, University of Utah
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: DOD02
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Knee Pain Chronic
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Our design is a sequential multiple randomization (SMART) study design with 2 treatment phases with a possibility of 2 randomizations per participant.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Brief mindfulness followed by brief mindfulness for non-responders (Experimental): 1 session of brief mindfulness, plus standard of care. At the one-month post-surgical follow-up, non-responders will receive another single session of brief mindfulness. Responders will continue to receive standard of care.
  Interventions: Behavioral: Brief mindfulness
- Standard care followed by brief mindfulness for non-responders (Experimental): Patients will attend a 2-hour preoperative class involving pain coping education and are offered prehabilitation services. At the one-month post-surgical follow-up, non-responders will receive one session of brief mindfulness. Responders will continue to receive standard of care.
  Interventions: Behavioral: Brief mindfulness; Other: Standard care
- Brief mindfulness followed by MORE for non-responders (Experimental): 1 session of brief mindfulness, plus standard of care. At the one-month post-surgical follow-up, non-responders will receive the 8 session MORE intervention. Responders will continue to receive standard of care.
  Interventions: Behavioral: Brief mindfulness; Behavioral: Mindfulness-Oriented Recovery Enhancement (MORE)
- Standard care followed by MORE for non-responders (Experimental): Patients will attend a 2-hour preoperative class involving pain coping education and are offered prehabilitation services. At the one-month post-surgical follow-up, non-responders will receive the 8 session MORE intervention. Responders will continue to receive standard of care.
  Interventions: Behavioral: Mindfulness-Oriented Recovery Enhancement (MORE); Other: Standard care

INTERVENTIONS:
Behavioral: Brief mindfulness — A 15-minute guided mindfulness practice that includes focused attention on breath and body sensations and open monitoring and acceptance of thoughts, emotions, and pain.
  Arms: Brief mindfulness followed by MORE for non-responders; Brief mindfulness followed by brief mindfulness for non-responders; Standard care followed by brief mindfulness for non-responders
Behavioral: Mindfulness-Oriented Recovery Enhancement (MORE) — An 8-session intervention. Sessions involve: 1) mindfulness training to reduce pain and increase self-regulation over opioid use, 2) cognitive reappraisal to decrease psychological distress, and 3) savoring to augment natural reward processing, positive emotion, and esprit de corps.
  Arms: Brief mindfulness followed by MORE for non-responders; Standard care followed by MORE for non-responders
Other: Standard care — Preoperative Standard Care. Patients will attend a 2-hour preoperative class involving pain coping education and are offered prehabilitation services. Postoperative standard care includes (1) pain medications to minimize opioid use, including acetaminophen, lyrica, meloxicam/naproxen and celebrex, and (2) anticoagulants for 3-6 weeks postoperatively, as well as (3) ambulatory care with assistive devices 1-6 weeks after surgery. Patients see their surgeon postoperatively 2-6 weeks after surgery, 3-6 months, and yearly.
  Arms: Standard care followed by MORE for non-responders; Standard care followed by brief mindfulness for non-responders

SUMMARY:
The overarching objective of this proposal is to conduct a multi-site Sequential Multiple Assignment Randomized Trial (SMART) across multiple Military Health System (MHS) sites to optimize the sequencing and integration of two intervention strategies in total knee arthoplasty (TKA) patients: a single-session mindfulness-based intervention (MBI) and an intensive 8-week MBI-Mindfulness-Oriented Recovery Enhancement (MORE) designed to simultaneously reduce prolonged pain and chronic opioid use by enhancing self-regulation. Aim 1: Evaluate the extent to which a brief preoperative MBI improves TKA patients' postoperative musculoskeletal health and reduces chronic opioid use. Aim 2: Evaluate the extent to which an intensive MBI (MORE) improves musculoskeletal health and reduces chronic opioid use among patients non-responsive to preoperative intervention. Aim 3: (A) Determine patient baseline characteristics that moderate MBI treatment responses. (B) Quantify the degree to which the impact of Phase 1 and 2 MBIs on musculoskeletal health and opioid dose are mediated by changes in mechanistic autonomic marker of self-regulation: heart-rate variability (HRV).

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo unilateral total TKA at one of the study sites
* TRICARE beneficiary
* Facility with the English language that is adequate to complete study procedures.

Exclusion Criteria:

* Cognitive impairment preventing completion of study procedures,
* Formal mindfulness training (e.g., MBSR, MBCT)
* Severe, active suicidality
* Contralateral TKA in the past 3 months or planned contralateral TKA during the study
* Current cancer diagnoses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster (WOMAC) Universities Osteoarthritis Index | Baseline to 9 months
  Western Ontario and McMaster (WOMAC) Universities Osteoarthritis Index (min 0, max 240, with higher scores indicating worse osteoarthritis).

SECONDARY OUTCOMES:
Opioid use | Baseline to 9 months
  Opioid use will be assessed by triangulating EHR data from the pharmacy data transaction service (PDTS) with real-time self-reports using a smartphone-enabled daily diary and retrospective reports with the validated Timeline Followback procedure.
Distress | Baseline to 9 months
  Depression Anxiety and Stress Scale (range from 0 to 63, higher scores indicating worse distress)
Defense and Veterans Pain Rating Scale | Baseline to 9 months
  Defense and Veterans Pain Rating Scale, a numeric rating scale enhanced by word descriptors, color coding, and pictorial facial expressions matched to pain levels (0 to 10, higher scores indicating worse pain)
Opioid misuse | Baseline to 9 months
  Current Opioid Misuse Measure (0 to 68, higher scores indicating higher opioid misuse)
Health-related quality of life | Baseline to 9 months
  EuroQol EQ-5D (1 to 5, with higher scores indicating lower quality of life)

OTHER OUTCOMES:
Perceived ability to return to duty | Baseline to 9 months
  3 questions assessing a service member's self-perceived ability to perform military related tasks (pass a required semi-annual physical fitness test, operate under full combat load, and % mission capability)
Pleasant body sensations | Baseline to 9 months
  Pleasant sensation ratio as measured by Sensation Manikin, a measure comprised of a visual body map to demonstrate the location and distribution of sensations.
Self-transcendence | Baseline to 9 months
  Self-transcendence measured by Nondual Awareness Dimensional Assessment, with higher scores indicating higher self-transcendence (min 13, max 65)
Positive affect | Baseline to 9 months
  Positive affect measured by numeric rating scale, with higher scores indicating higher positive affect (min 0, max 10)
Mindful reinterpretation of pain sensations | Baseline to 9 months
  Mindful reinterpretation of pain sensations (min 0, max 54, with higher scores indicating greater mindful reappraisal of pain)
Heart rate variability | Baseline,1 month, 3 months
  Change in HRV (mindfulness - resting baseline, higher values representing more HRV)
Trait mindfulness | Baseline to 9 months
  Five Facet Mindfulness Questionnaire (min 39, max 195, higher scores indicating greater mindfulness)
Cognitive reappraisal | Baseline to 9 months
  Reappraisal subscale of the Cognitive Emotion Regulation Questionnaire (min 4, max 20, higher scores indicating more reappraisal)
Savoring natural rewards | Baseline to 9 months
  Brief savoring inventory (min 4, max 20, higher scores indicating more savoring)

CONTACTS AND LOCATIONS:
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided